CLINICAL TRIAL: NCT00675714
Title: Assessment of the Treatment of the Severely Burned With Anabolic Agents on Clinical Outcomes, Recovery and Rehabilitation
Brief Title: Assessment of the Treatment of Severely Burned With Anabolic Agents on Clinical Outcomes, Recovery and Rehabilitation
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: At the request of the study site, this study has been closed and access to study-related data is unavailable. We are unable to submit the results-data.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency); National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-157; NIDILRR 90DP0043-03-00; P50GM060338 (NIH)
Record Dates: First submitted 2007-12-26; First posted 2008-05-12 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2018-08

CONDITIONS: Burns
Keywords: anabolic agents; exercise
MeSH Terms: conditions — Burns; Motor Activity | interventions — Absorptiometry, Photon; High-Energy Shock Waves; Magnetic Resonance Spectroscopy; Human Growth Hormone; Growth Hormone; Ketoconazole; Itraconazole; Fluconazole; Oxandrolone; Testosterone; Nandrolone; Propranolol; Metoprolol; Exercise; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- 1 (Experimental): Humatrope subcutaneous(SQ) 0.05-0.2 mg/kg/day for up to 2 years post burn
  Interventions: Procedure: Stable Isotope Infusion Study; Procedure: Collection of blood and tissues; Procedure: Radiology testing: Dual-energy X-ray absorptiometry (DEXA), ultrasound, MRI; Drug: Humatrope
- 2 (Experimental): Ketoconazole by mouth (PO) given twice a day throughout hospitalization for up to 2 years post burn
  Interventions: Procedure: Stable Isotope Infusion Study; Procedure: Collection of blood and tissues; Procedure: Radiology testing: Dual-energy X-ray absorptiometry (DEXA), ultrasound, MRI; Drug: Ketoconazole
- 3 (Experimental): Oxandrolone PO given daily throughout hospitalization for up to 2 years post burn
  Interventions: Procedure: Stable Isotope Infusion Study; Procedure: Collection of blood and tissues; Procedure: Radiology testing: Dual-energy X-ray absorptiometry (DEXA), ultrasound, MRI; Drug: Oxandrolone
- 4 (Experimental): Propranolol PO given daily throughout hospitalization for up to 2 years post burn
  Interventions: Procedure: Stable Isotope Infusion Study; Procedure: Collection of blood and tissues; Procedure: Radiology testing: Dual-energy X-ray absorptiometry (DEXA), ultrasound, MRI; Drug: Propranolol
- 5 (Experimental): Oxandrolone and propranolol PO to be given daily for up to 2 years post burn
  Interventions: Procedure: Stable Isotope Infusion Study; Procedure: Collection of blood and tissues; Procedure: Radiology testing: Dual-energy X-ray absorptiometry (DEXA), ultrasound, MRI; Drug: Oxandrolone and propranolol combined
- 6 (Experimental): Humatrope SQ and Propranolol PO to be given daily for up to 2 years post burn
  Interventions: Procedure: Stable Isotope Infusion Study; Procedure: Collection of blood and tissues; Procedure: Radiology testing: Dual-energy X-ray absorptiometry (DEXA), ultrasound, MRI; Drug: Humatrope and propranolol combined
- 7 (Placebo Comparator): Placebo PO to be given for up to 2 years post burn
  Interventions: Procedure: Stable Isotope Infusion Study; Procedure: Collection of blood and tissues; Procedure: Radiology testing: Dual-energy X-ray absorptiometry (DEXA), ultrasound, MRI; Drug: Placebo
- 8 (Experimental): Exercise--hospital supervised intensive exercise program
  Interventions: Procedure: Stable Isotope Infusion Study; Procedure: Collection of blood and tissues; Procedure: Radiology testing: Dual-energy X-ray absorptiometry (DEXA), ultrasound, MRI; Behavioral: Exercise--Hospital supervised intensive exercise program
- 9 (Experimental): Exercise--home or community based exercise program
  Interventions: Procedure: Stable Isotope Infusion Study; Procedure: Collection of blood and tissues; Procedure: Radiology testing: Dual-energy X-ray absorptiometry (DEXA), ultrasound, MRI; Behavioral: Home exercise program

INTERVENTIONS:
Procedure: Stable Isotope Infusion Study — 1-8 hour stable isotope infusion study to be done following each surgery. Tagged isotopes to assess uptake into blood and tissues.
Procedure: Collection of blood and tissues — Blood draw with each stable isotope infusion study and weekly Tissue biopsy: skin, fat, muscle at stable isotope infusion study
Procedure: Radiology testing: Dual-energy X-ray absorptiometry (DEXA), ultrasound, MRI — Testing to be done following every stable isotope infusion study to measure muscle, fat and bone tissues.
Drug: Humatrope — Humatrope (Growth Hormone) dose:0.05mg - 0.2mg/kg/day SQ daily for up to 2 years post burn injury.
  Other Names: recombinant human growth hormone; Growth Hormone
  Arms: 1
Drug: Ketoconazole — Ketoconazole administration (or other glucocorticoid blocker--itraconazole or fluconazole) PO daily for up to 2 years post burn injury
  Other Names: itraconazole; fluconazole
  Arms: 2
Drug: Oxandrolone — oxandrolone (or other anabolic steroid-testosterone or nandrolone) daily for up to 2 years post burn injury
  Other Names: testosterone; nandrolone
  Arms: 3
Drug: Propranolol — Propranolol (or other beta adrenergic blocker--metoprolol, inderol), PO administration daily for up to 2 years post burn injury.
  Other Names: metoprolol; inderol
  Arms: 4
Drug: Oxandrolone and propranolol combined — Daily administration of oxandrolone and propranolol to be given for up to 2 years post burn injury.
  Other Names: testosterone; nandrolone; inderol; metoprolol
  Arms: 5
Drug: Humatrope and propranolol combined — Humatrope (growth hormone) and propranolol administration daily for up to 2 years post burn injury.
  Other Names: recombinant human growth hormone; Growth Hormone; inderol; metoprolol
  Arms: 6
Drug: Placebo — placebo to be given once a day for up to two years post burn injury.
  Other Names: control
  Arms: 7
Behavioral: Exercise--Hospital supervised intensive exercise program — intensive exercise program supervised by trained personnel in the hospital environment for six up to twelve week program.
  Other Names: exercise; intensive exercise; aerobic exercise; exercise rehabilitation program; hospital based exercise
  Arms: 8
Behavioral: Home exercise program — Home intensive exercise program: training occurs in hospital then patient sent home to continue exercise program for six weeks and up to 12 weeks at home.
  Other Names: Home exercise; intensive exercise; exercise rehabilitation
  Arms: 9

SUMMARY:
The purpose of the program is to study and characterize the outcome of burn injury with particular attention to improving the rehabilitation of burn survivors, including children. Various agents are assessed for effectiveness on long term burn outcome, such as growth hormone, oxandrolone, propranolol,ketoconazole, inhospital exercise and home exercise.

DETAILED DESCRIPTION:
The University of Texas Medical Branch(UTMB) project improves outcomes for severely burned children by instituting and evaluating two modifications to traditional rehabilitation: (1) an intensive rehabilitation program including active resistance exercise; (2) long term administration of anabolic agents.

Effectiveness is assessed by comparison with functional outcomes achieved in traditional outpatient rehabilitation programs. Results indicate improvement in strength, endurance and bone density with these modifications. The project also maintains a longitudinal database that includes measures of cardiopulmonary function, growth and maturation, bone density, range of motion, and psychosocial adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Burn 30% Total Body Surface Area (TBSA) or greater
* Ages 0-80 yrs
* Negative pregnancy test
* Informed consent

Exclusion Criteria:

* Untreated malignancy, known history of AIDS, Aids Related Complex, HIV
* Recent history of myocardial infarction (6 wks)
* Tuberculosis, arthritis, cirrhosis, hyperlipidemia, bone or endocrine diseases, autoimmune diseases
* Chronic glucocorticoid or non steroidal anti inflammatory drug therapy
* Diabetes mellitus prior to burn injury
* Renal insufficiency (defined by creatinine >3.0 mg/dl)
* Hepatic disease (bilirubin > 3.0 mg/dl)

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1126 (Actual)
Dates: Start 2004-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Measures of muscle wasting, weakness, immunosuppression chronic bone loss and decreased growth with increases in metabolic, hemodynamic, inflammatory and scarring responses. | Admission to burn unit and up to 2 years post burn and yearly after that
  Dual Energy X-Ray Absorptiometry measurements will be utilized to measure muscle wasting

CONTACTS AND LOCATIONS:
Overall Officials: David N Herndon, MD, Study Director — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alloju SM, Herndon DN, McEntire SJ, Suman OE. Assessment of muscle function in severely burned children. Burns. 2008 Jun;34(4):452-9. doi: 10.1016/j.burns.2007.10.006. Epub 2008 Feb 20. PMID 18243565
- [Derived] Guillory AN, Herndon DN, Silva MB 3rd, Andersen CR, Suman OE, Finnerty CC. Oxandrolone Coadministration Does Not Alter Plasma Propranolol Concentrations in Severely Burned Pediatric Patients. J Burn Care Res. 2017 Jul/Aug;38(4):243-250. doi: 10.1097/BCR.0000000000000494. PMID 28240622
- [Derived] Herndon DN, Voigt CD, Capek KD, Wurzer P, Guillory A, Kline A, Andersen CR, Klein GL, Tompkins RG, Suman OE, Finnerty CC, Meyer WJ, Sousse LE. Reversal of Growth Arrest With the Combined Administration of Oxandrolone and Propranolol in Severely Burned Children. Ann Surg. 2016 Sep;264(3):421-8. doi: 10.1097/SLA.0000000000001844. PMID 27433905
- [Derived] Sousse LE, Herndon DN, Mlcak RP, Lee JO, Andersen CR, Zovath AJ, Finnerty CC, Suman OE. Long-Term Administration of Oxandrolone Improves Lung Function in Pediatric Burned Patients. J Burn Care Res. 2016 Sep-Oct;37(5):273-7. doi: 10.1097/BCR.0000000000000356. PMID 27171844
- [Derived] Diaz EC, Herndon DN, Lee J, Porter C, Cotter M, Suman OE, Sidossis LS, Borsheim E. Predictors of muscle protein synthesis after severe pediatric burns. J Trauma Acute Care Surg. 2015 Apr;78(4):816-22. doi: 10.1097/TA.0000000000000594. PMID 25807408
- [Derived] Kraft R, Herndon DN, Finnerty CC, Cox RA, Song J, Jeschke MG. Predictive Value of IL-8 for Sepsis and Severe Infections After Burn Injury: A Clinical Study. Shock. 2015 Mar;43(3):222-7. doi: 10.1097/SHK.0000000000000294. PMID 25514427
- [Derived] Patel P, Sallam HS, Ali A, Chandalia M, Suman O, Finnerty CC, Herndon DN, Abate N. Changes in fat distribution in children following severe burn injury. Metab Syndr Relat Disord. 2014 Dec;12(10):523-6. doi: 10.1089/met.2014.0098. Epub 2014 Sep 11. PMID 25211297
- [Derived] Chondronikola M, Meyer WJ, Sidossis LS, Ojeda S, Huddleston J, Stevens P, Borsheim E, Suman OE, Finnerty CC, Herndon DN. Predictors of insulin resistance in pediatric burn injury survivors 24 to 36 months postburn. J Burn Care Res. 2014 Sep-Oct;35(5):409-15. doi: 10.1097/BCR.0000000000000017. PMID 24918945
- [Derived] Hardee JP, Porter C, Sidossis LS, Borsheim E, Carson JA, Herndon DN, Suman OE. Early rehabilitative exercise training in the recovery from pediatric burn. Med Sci Sports Exerc. 2014 Sep;46(9):1710-6. doi: 10.1249/MSS.0000000000000296. PMID 24824900
- [Derived] Finnerty CC, Ali A, McLean J, Benjamin N, Clayton RP, Andersen CR, Mlcak RP, Suman OE, Meyer W, Herndon DN. Impact of stress-induced diabetes on outcomes in severely burned children. J Am Coll Surg. 2014 Apr;218(4):783-95. doi: 10.1016/j.jamcollsurg.2014.01.038. Epub 2014 Jan 24. PMID 24655871
- [Derived] Finnerty CC, Herndon DN. Is propranolol of benefit in pediatric burn patients? Adv Surg. 2013;47:177-97. doi: 10.1016/j.yasu.2013.02.001. No abstract available. PMID 24298851
- [Derived] Finnerty CC, Mabvuure NT, Ali A, Kozar RA, Herndon DN. The surgically induced stress response. JPEN J Parenter Enteral Nutr. 2013 Sep;37(5 Suppl):21S-9S. doi: 10.1177/0148607113496117. PMID 24009246
- [Derived] Ray S, Ju X, Sun H, Finnerty CC, Herndon DN, Brasier AR. The IL-6 trans-signaling-STAT3 pathway mediates ECM and cellular proliferation in fibroblasts from hypertrophic scar. J Invest Dermatol. 2013 May;133(5):1212-20. doi: 10.1038/jid.2012.499. Epub 2013 Jan 10. PMID 23303450
- [Derived] Kraft R, Herndon DN, Finnerty CC, Hiyama Y, Jeschke MG. Association of postburn fatty acids and triglycerides with clinical outcome in severely burned children. J Clin Endocrinol Metab. 2013 Jan;98(1):314-21. doi: 10.1210/jc.2012-2599. Epub 2012 Nov 12. PMID 23150682
- [Derived] Herndon DN, Rodriguez NA, Diaz EC, Hegde S, Jennings K, Mlcak RP, Suri JS, Lee JO, Williams FN, Meyer W, Suman OE, Barrow RE, Jeschke MG, Finnerty CC. Long-term propranolol use in severely burned pediatric patients: a randomized controlled study. Ann Surg. 2012 Sep;256(3):402-11. doi: 10.1097/SLA.0b013e318265427e. PMID 22895351
- [Derived] Jeschke MG, Williams FN, Finnerty CC, Rodriguez NA, Kulp GA, Ferrando A, Norbury WB, Suman OE, Kraft R, Branski LK, Al-mousawi AM, Herndon DN. The effect of ketoconazole on post-burn inflammation, hypermetabolism and clinical outcomes. PLoS One. 2012;7(5):e35465. doi: 10.1371/journal.pone.0035465. Epub 2012 May 11. PMID 22606232
- [Derived] Porro LJ, Herndon DN, Rodriguez NA, Jennings K, Klein GL, Mlcak RP, Meyer WJ, Lee JO, Suman OE, Finnerty CC. Five-year outcomes after oxandrolone administration in severely burned children: a randomized clinical trial of safety and efficacy. J Am Coll Surg. 2012 Apr;214(4):489-502; discussion 502-4. doi: 10.1016/j.jamcollsurg.2011.12.038. PMID 22463890
- [Derived] Traber MG, Leonard SW, Traber DL, Traber LD, Gallagher J, Bobe G, Jeschke MG, Finnerty CC, Herndon D. alpha-Tocopherol adipose tissue stores are depleted after burn injury in pediatric patients. Am J Clin Nutr. 2010 Dec;92(6):1378-84. doi: 10.3945/ajcn.2010.30017. Epub 2010 Sep 29. PMID 20881067
- [Derived] Branski LK, Herndon DN, Barrow RE, Kulp GA, Klein GL, Suman OE, Przkora R, Meyer W 3rd, Huang T, Lee JO, Chinkes DL, Mlcak RP, Jeschke MG. Randomized controlled trial to determine the efficacy of long-term growth hormone treatment in severely burned children. Ann Surg. 2009 Oct;250(4):514-23. doi: 10.1097/SLA.0b013e3181b8f9ca. PMID 19734776
- See also: University of Texas web page to describe funded program — http://www.utmb.edu/sbhnidrr/
- See also: burn care web site includes information on funded grant project — http://www.totalburncare.com